CLINICAL TRIAL: NCT03678467
Title: An Open-Label, First-in-Human, Single Intervention Study for Evaluation of EpiBone-CMF Engineered Living Bone Graft for Mandibular Ramus Reconstruction
Brief Title: Evaluation of EpiBone-CMF for Mandibular Ramus Reconstruction
Acronym: EB-CMF
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Epibone, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EB-CMF-02
Record Dates: First submitted 2018-09-12; First posted 2018-09-19 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Mandible Tumor; Mandibular Injuries; Mandible; Deformity
Keywords: tissue engineering, tissue engineered product, mesenchymal stem cells
MeSH Terms: conditions — Mandibular Neoplasms; Mandibular Injuries; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- EB-CMF Implant (Experimental): Subject receiving EB-CMF implant
  Interventions: Combination Product: EB-CMF

INTERVENTIONS:
Combination Product: EB-CMF — Autologous, anatomically shaped bone graft

SUMMARY:
EpiBone-Craniomaxillofacial (EB-CMF) is an autologous, anatomically shaped bone graft created specifically for the patient's defect, using the patients own adipose-derived mesenchymal stem cells. This first in human trial is designed specifically to assess the safety of EB-CMF clinically. Although secondary measures of graft efficacy are being assessed, the primary focus will be on Adverse Events stemming from graft implantation.

ELIGIBILITY:
Inclusion Criteria

1. Patients must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
2. Stable mandibular ramus injury or defect due to trauma, disease, or congenital defects.
3. Medical history must be verified by either a personal physician or medical practitioner as appropriate.
4. Patient determined by the Investigator to be a suitable candidate by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac evaluation.
5. A female patient is eligible to participate if she is not pregnant (see Appendix 6), not breastfeeding, and at least 1 of the following conditions applies:

   1. A woman of nonchildbearing potential (WONCBP) as defined in Appendix 6. OR
   2. A woman of childbearing potential (WOCBP) who agrees to follow the contraceptive guidance in Appendix 6 for at least 1 month prior to surgery, during the treatment period, and until 12 weeks after completion of the study.
6. Patient must be available at the study center for all specified assessments throughout the study duration.
7. Patients whose clinical laboratory test results are within the reference range for healthy individuals, or where outside the reference range is judged as not clinically relevant by the Investigator.
8. All patients are required to give written informed consent as described in Appendix 2, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol, and in accordance with the Declaration of Helsinki, before enrollment. Patients must provide written informed consent and authorization for use and disclosure of protected health information.
9. A healthy condyle which can be plated with titanium plates and screws.
10. A mandibular continuity ramus defect which starts below the sigmoid notch and extends only as far as but not including the angle.

Exclusion Criteria

1. Uncontrolled alcohol, tobacco, or substance abuse within 6 months prior to implantation.
2. Mandibular ramus defects with open wounds.
3. Defects > 15 cc in volume.
4. Defects > 6 cm in diameter.
5. Systemic disease that would render the fat harvest and product implantation, along with associated anesthesia, unsafe to the patient.
6. Patient has any underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would impact patient safety or interfere with the integrity of the study data.
7. Active uncontrolled infection or malignancy. Patients will be allowed to undergo rescreening once, after the infection is cleared, if they are willing to do so.
8. Patients with signs and symptoms of infection between Screening and up to the surgical implantation.
9. Radiation therapy < 6 months prior to the surgical implantation.
10. Need for soft tissue reconstruction (flap, skin graft, etc).
11. Conditions that may impact the success of the surgical implantation or increase the risk of postoperative complications, including inherited coagulopathies like hemophilia, Von Willebrand's disease, protein C and S deficiency, thrombocythemias, thallassemias, sickle cell disease, etc.
12. Conditions that may impact functional outcomes, including uncontrolled diabetes, osteoporosis, rare disorders of bone healing like osteopetrosis, or any other metabolic bone disease.
13. Increased alkaline phosphatase (to exclude Paget's disease), increased serum calcium (to exclude hyperparathyroidism), or Vitamin D deficiency, at Screening, confirmed by a repeat test.
14. Oral bisphosphonate < 12 weeks, intravenous bisphosphonate < 12 months prior to Screening or use of systemic steroids or anabolic agents (e.g. teriparatide) for osteoporosis treatment.
15. Patients with inadequate donor sites for lipoaspirate of adipose tissue.
16. Mixed connective tissue diseases and collagen diseases which can result in poor wound healing after surgery.
17. Patients considered unsuitable per the consulted surgeon.
18. Patient has any of the following conditions as identified by medical history:

    1. Human immunodeficiency virus (active or seropositive).
    2. Active tuberculosis.
    3. Active hepatitis B infection.
    4. Hepatitis C.
    5. Viral encephalitis.
    6. Toxoplasmosis. In case of doubt regarding mentioned conditions based on the physical examination or other signs or symptoms present at Screening, the patient will be asked to consent to additional testing to rule out such conditions or the patient must be excluded from the study.
19. Donation of blood and blood products is not permitted from Screening and for at least 3 months after the surgical implantation.
20. Patient participated in another clinical study of an investigational drug within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to the surgical implantation or is currently participating in another clinical study of an investigational drug or intending to participate in another clinical study of an investigational drug before completion of all scheduled evaluations in this clinical study.
21. Patients who, in the opinion of the Investigator, are not likely to complete the study for whatever reason.
22. The Investigator or any sub-investigator, research assistant, surgeon, study coordinator, or other staff directly involved in the conduct of the clinical study or any of their relatives.
23. Hypersensitivity to any product of bovine origin.
24. Hypersensitivity to gentamicin or other aminoglycosides.
25. Post-menopausal women who have an abnormally low bone mineral density or have not tested for bone mineral density.
26. Patients with discontinuity defects of the ramus.
27. Patients with a history of malignant cancer.
28. Hypersensitivity or allergy to epinephrine or other drugs commonly used during surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | 12 months
  To assess the safety of EB-CMF for up to 12 months post surgery in subjects with recent or remote mandibular ramus defects requiring up to a 15 cc graft reconstruction.

SECONDARY OUTCOMES:
Bone regeneration as assessed by high-resolution CT scans | 12 months
  To assess the efficacy of the EpiBone-CMF graft for up to 12 months post-surgery in subjects with recent or remote mandibular ramus defects requiring up to a 15 cc graft reconstruction. Bone regeneration as assessed by high-resolution CT scans for up to 12 months post-surgery.
Quality of life as measured by the Glasgow Benefit Inventory | 12 months
  To assess the changes in quality of life for up to 12 months post-surgery in patients as measured by the Glasgow Benefit Inventory.
Quality of life as measured by SF-12 | 12 months
  To assess the changes in quality of life for up to 12 months post-surgery in patients as measured by SF-12.

OTHER OUTCOMES:
Observational assessment of bone regeneration by high-resolution CT scan | 10 Years
  Yearly observation of bone regeneration by high-resolution CT scan until the subject withdraws from the study or termination of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Gastman, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - VA Healthcare System, San Francisco, San Francisco, California
  - Cleveland Clinic, Cleveland, Ohio
  - UT Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bhumiratana S, Bernhard JC, Alfi DM, Yeager K, Eton RE, Bova J, Shah F, Gimble JM, Lopez MJ, Eisig SB, Vunjak-Novakovic G. Tissue-engineered autologous grafts for facial bone reconstruction. Sci Transl Med. 2016 Jun 15;8(343):343ra83. doi: 10.1126/scitranslmed.aad5904. PMID 27306665
- [Background] Bhumiratana S, Vunjak-Novakovic G. Concise review: personalized human bone grafts for reconstructing head and face. Stem Cells Transl Med. 2012 Jan;1(1):64-9. doi: 10.5966/sctm.2011-0020. Epub 2011 Dec 7. PMID 23197642
- [Background] Grayson WL, Marolt D, Bhumiratana S, Frohlich M, Guo XE, Vunjak-Novakovic G. Optimizing the medium perfusion rate in bone tissue engineering bioreactors. Biotechnol Bioeng. 2011 May;108(5):1159-70. doi: 10.1002/bit.23024. Epub 2010 Dec 22. PMID 21449028
- [Background] Grayson WL, Bhumiratana S, Cannizzaro C, Vunjak-Novakovic G. Bioreactor cultivation of functional bone grafts. Methods Mol Biol. 2011;698:231-41. doi: 10.1007/978-1-60761-999-4_18. PMID 21431523
- See also: EpiBone, Inc. — http://www.epibone.com